CLINICAL TRIAL: NCT01412489
Title: Prevention of Postsurgical Uterine Synechia With HyalobarrierR Gel Endo in Hysteroscopic Myomectomy : a Prospective Multicenter Study
Brief Title: Intrauterine Adhesion Rate After Hysteroscopic Myomectomy and Application of HYALOBARRIER Gel
Acronym: HYGEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: K 100801
Record Dates: First submitted 2011-05-16; First posted 2011-08-09 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Myoma
Keywords: Uterine synechiae; HyalobarrierR Gel Endo; Operative hysteroscopy; submucous myoma
MeSH Terms: conditions — Myoma; Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): For each patient, the HYALOBARRIER Gel was introduced into the uterine cavity with the canula after hysteroscopic myomectomy procedure
  Interventions: Device: HYALOBARRIER Gel

INTERVENTIONS:
Device: HYALOBARRIER Gel — For each patient, the HYALOBARRIER Gel was introduced into the uterine cavity with the canula after hysteroscopic myomectomy procedure

SUMMARY:
The purpose of this study is to evaluate the intrauterine adhesion rate after the application of HYALOBARRIER Gel at the end of hysteroscopic myomectomy. Secondary endpoints were tolerance and side effect and subsequent fertility.

DETAILED DESCRIPTION:
Hysteroscopic myomectomy is the referent surgical treatment for submucous myoma. But intrauterine adhesion rate was evaluated about 7 to 15% after this procedure. The investigators hypothetically believe that application of HYALOBARRIER Gel at the end of the procedure, could be reduce the mean intrauterine rate to 50%. Thus, the investigators performed a multicenter (n = 20) prospective study non randomized in 220 patients with submucous myoma < 3 cm of diameter, evaluated by preoperative ultrasound. The investigators prefer this study design, because the principal reason is the number of enrolled patient were more 200 patients in each group with a double blind randomized study. Now, in all patients, after hysteroscopic myomectomy which performed with a same technique in each center (bipolar coagulation and physiologic serum), a diagnostic hysteroscopy was performed at 2 month to determinate the existence of intrauterine adhesion. Secondary end points were in this study the tolerance and side effects of HYALOBARRIER Gel and the subsequent fertility at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 aged-patients
* hysteroscopic diagnosis of one submucous myoma with less than 3cm diameter requiring operative hysteroscopy with saline type 0, 1 or 2
* negative plasmatic βHCG test
* non opposition
* patients with social security

Exclusion Criteria:

* multiple submucous myomas type 0, 1 or 2
* presurgical embolization
* presurgical impregnation with GnRH agonist
* coagulative disorders
* malignancies
* uncontrolled diabetes
* operative hysteroscopy with glycine
* known hypersensitivity to HyalobarrierR Gel Endo
* infection of the surgical area concerned

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The formation of postsurgical uterine synechiae rate with HyalobarrierR Gel Endo in hysteroscopic myomectomy | between 4 and 8 weeks after initial hysteroscopic myomectomy

SECONDARY OUTCOMES:
the number of participants with adverse events as a measure of safety and tolerability during the time of the study | 2 years
Postsurgical fertility with evaluation of number of participants who became pregnant after surgery, spontaneously and/or after assisted reproductive technologies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Benifla, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de Gynecologie-Obstetrique, Hopital Lariboisière, Paris, France